CLINICAL TRIAL: NCT00068822
Title: Investigational Vertebroplasty Efficacy and Safety Trial (INVEST)
Brief Title: Vertebroplasty for the Treatment of Fractures Due to Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: David F. Kallmes, MD (PI), Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1912-03; R01AR049373 (NIH); NIAMS-096; UL1RR025014 (NIH)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Spinal Fractures; Osteoporosis
Keywords: Vertebroplasty; Crushed Vertebrae; Back Pain; Structurally Unstable Vertebrae; polymethylmethacrylate; INVEST; PMMA; RDQ
MeSH Terms: conditions — Spinal Fractures; Osteoporosis; Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vertebroplasty (Experimental): Participants will receive percutaneous vertebroplasty
  Interventions: Device: Percutaneous vertebroplasty
- Control Group (Placebo Comparator): Participants will receive sham vertebroplasty without PMMA
  Interventions: Procedure: Sham vertebroplasty

INTERVENTIONS:
Device: Percutaneous vertebroplasty — Placement of polymethylmethacrylate (PMMA) into vertebral compression fracture
  Arms: Vertebroplasty
Procedure: Sham vertebroplasty — Participants, following local anesthesia with lidocaine and bupivacaine, were given verbal and physical cues such as pressure on the back, but the needle was not placed.
  Arms: Control Group

SUMMARY:
Vertebroplasty is a procedure used to stabilize broken vertebrae, the bones that form the spine. This study will evaluate the effectiveness of vertebroplasty for the treatment of fractures due to osteoporosis.

DETAILED DESCRIPTION:
Spontaneous, atraumatic compression fractures due to osteoporosis occur in more than 700,000 patients per year. Pain associated with these fractures may be excruciating, but before the advent of percutaneous vertebroplasty, treatment options were limited. Analgesic medications, bed rest, and bracing have been the mainstays of treatment, but each of these therapies has substantial limitations.

Because of the dearth of viable treatment options for osteoporotic vertebral compression fractures, the practice of percutaneous vertebroplasty, which involves injection of polymethylmethacrylate (medical cement) into the fractured vertebra, has disseminated rapidly. However, evidence for the efficacy of percutaneous vertebroplasty is currently limited to uncontrolled, nonblinded, small case studies. Even though high rates of success are reported, with up to 90% of patients achieving substantial pain relief, these case studies have not accounted for numerous important potential biases, including the natural tendency for compression fractures to heal spontaneously, regression toward the mean (wherein patients seek medical attention when pain is maximum), and the placebo effect. This study will examine the clinical efficacy of percutaneous vertebroplasty for treatment of painful osteoporotic vertebral compression fractures.

Participants in this study will be randomly assigned to receive either percutaneous vertebroplasty or a sham procedure (placebo control group). Participants may have up to 2 spinal levels treated. Participants will be enrolled in the study for 1 year and will have study visits at entry and Months 1 and 12. There will also be phone visits at Days 1, 2, 3, and 14 and Months 3 and 6. After Month 1, crossover from the placebo group to the vertebroplasty group will be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed osteoporosis or osteopenia by a referring physician and/or medical history and physical exam OR osteopenia on plain film
* Vertebral compression fracture in vertebrae T4 through L5, of less than 1 year old
* Pain not responsive to standard medical therapy
* Current rating for pain intensity of at least 3 on a scale of 0 to 10

Exclusion Criteria:

* Evidence or suspicion of malignant tumor or spinal canal compromise
* Concomitant hip fracture
* Local or systemic infection
* Uncorrectable bleeding diatheses
* Surgery within the previous 60 days
* Lack of access to telephone
* Inability to communicate in English
* Dementia
* Pregnancy
* Abnormal renal function or anticipated venography
* Conscious sedation is contraindicated for subject

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2003-04; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F. Kallmes, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Kallmes DF, Jensen ME. Percutaneous vertebroplasty. Radiology. 2003 Oct;229(1):27-36. doi: 10.1148/radiol.2291020222. PMID 14519867
- [Result] Kallmes DF, Comstock BA, Heagerty PJ, Turner JA, Wilson DJ, Diamond TH, Edwards R, Gray LA, Stout L, Owen S, Hollingworth W, Ghdoke B, Annesley-Williams DJ, Ralston SH, Jarvik JG. A randomized trial of vertebroplasty for osteoporotic spinal fractures. N Engl J Med. 2009 Aug 6;361(6):569-79. doi: 10.1056/NEJMoa0900563. PMID 19657122
- [Derived] Comstock BA, Sitlani CM, Jarvik JG, Heagerty PJ, Turner JA, Kallmes DF. Investigational vertebroplasty safety and efficacy trial (INVEST): patient-reported outcomes through 1 year. Radiology. 2013 Oct;269(1):224-31. doi: 10.1148/radiol.13120821. Epub 2013 May 21. PMID 23696683

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at five centers in the U.S., five centers in the United Kingdom and one center in Australia.
Groups:
- Vertebroplasty, Then Control: Participants randomized to receive percutaneous vertebroplasty first (placement of polymethylmethacrylate [PMMA] into vertebral compression fracture). At Month 1 or Month 3 if participants did not get enough pain relief from the procedure, they could opt to crossover to the alternative Control procedure, Sham Vertebroplasty (partial vertebroplasty without PMMA in which participants were given verbal and physical cues such as pressure on the back, following local anesthesia with lidocaine and bupivacaine, but the needle was not placed.)
- Control, Then Vertebroplasty: Participants randomized to receive Control procedure, Sham Vertebroplasty first (Partial vertebroplasty without PMMA in which participants were given verbal and physical cues such as pressure on the back, following local anesthesia with lidocaine and bupivacaine, but the needle was not placed.) At Month 1 or Month 3 if participants did not get enough pain relief from the procedure, they could opt to crossover to the alternative percutaneous vertebroplasty (placement of polymethylmethacrylate [PMMA] into vertebral compression fracture).
Period: First Randomized Intervention
Arm/Group | Vertebroplasty, Then Control | Control, Then Vertebroplasty
Started | 68 | 63
Completed | 67 | 61
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Period: Optional Crossover Intervention
Arm/Group | Vertebroplasty, Then Control | Control, Then Vertebroplasty
Started | 9 | 29
Crossover at Month 1 | 1 | 2
Crossover at Month 3 | 8 | 27
Completed | 9 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Participants will receive partial vertebroplasty without PMMA
- Total: Total of all reporting groups
Arm/Group | Vertebroplasty | Control Group | Total
Number analyzed (Participants) | 68 | 63 | 131
Age Continuous [Mean (Standard Deviation); unit: years] | 73.4 (9.4) | 74.3 (9.6) | 73.84 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 46 | 99
  Male | 15 | 17 | 32
Region of Enrollment [Number; unit: participants]
  United States | 29 | 28 | 57
  United Kingdom | 26 | 26 | 52
  Australia | 13 | 9 | 22
RDQ Score at baseline [Mean (Standard Deviation); unit: Units on a scale] — Scores on the Roland-Morris Disability Questionnaire (RDQ) range from 0-23, with higher scores indicating more severe disability
  Units on a scale | 16.6 (3.8) | 17.5 (4.1) | 17.05 (3.98)
Average pain intensity during past 24 hours at baseline [Mean (Standard Deviation); unit: Units on a scale] — The pain intensity rating ranges from 0 (no pain) to 10 (worst pain)
  Units on a scale | 6.9 (2.0) | 7.2 (1.8) | 7.02 (1.9)
SF-36 score; summary physical component at baseline [Mean (Standard Deviation); unit: Units on a scale] — Scores on the Medical Outcomes Study 36-Item Short-Form General Health Survey (SF-36), version 2. Subjects completed the SF-36 which consists of 8 sub-scales which are additionally summarized into 2 summary components (physical and mental). The subscales and the summary scales both range from 0 to 100, with (0 = worst imaginable, 100 = best imaginable).
  Units on a scale | 25.3 (7.8) | 25.3 (7.3) | 25.3 (7.55)
SF-36 score; summary mental component at baseline [Mean (Standard Deviation); unit: Units on a scale] — Scores on the Medical Outcomes Study 36-Item Short-Form General Health Survey (SF-36), version 2. Subjects completed the SF-36 which consists of 8 sub-scales which are additionally summarized into 2 summary components (physical and mental). The subscales and the summary scales both range from 0 to 100, with (0 = worst imaginable, 100 = best imaginable).
  Units on a scale | 44.8 (11.8) | 41.5 (14.1) | 43.21 (13.03)
Pain Frequency Index Score at baseline [Mean (Standard Deviation); unit: Units on a scale] — Scores on the Pain Frequency Index range from 0 to 4, with higher scores indicating more severe pain
  Units on a scale | 3.0 (0.8) | 3.1 (0.8) | 3.04 (0.8)
Pain Bothersome Index score at baseline [Mean (Standard Deviation); unit: Units on a scale] — Scores on the Pain Bothersome Index range from 0 to 4, with higher scores indicating more severe pain
  Units on a scale | 2.9 (0.7) | 3.1 (0.8) | 2.98 (0.75)
EQ-SD Score at baseline [Mean (Standard Deviation); unit: Units on a scale] — European Quality of Life - 5 Dimensions (EQ-SD) scale range from -0.1 to 1.0, with higher scores indicating a better quality of life.
  Units on a scale | 0.57 (0.18) | 0.54 (0.23) | 0.55 (0.20)
SOF-ADL Score at baseline [Mean (Standard Deviation); unit: Units on a scale] — Study of Osteoporotic Fractures - Activities of Daily Living (SOF-ADL) scale range from 0 to 18, with higher scores indicating more back-related disability
  Units on a scale | 10.0 (3.6) | 10.3 (2.8) | 10.14 (3.23)

OUTCOME MEASURES:

1. Primary Outcome: Back-specific Functional Status Using Roland-Morris Disability Questionnaire (RDQ) Scale at 1 Month
Description: Back-specific functional status using RDQ scale range from 0 (no pain) to 23, with higher scores indicating more severe disability.
Time Frame: 1 month after procedure
Population: 68 subjects were randomized to undergo vertebroplasty and 63 to undergo the control intervention. All underwent the assigned intervention. One subject in the vertebroplasty group and two subjects in the control group were lost to follow-up before 1 month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vertebroplasty | Control Group
Number analyzed (Participants) | 67 | 61
units on a scale | 12.0 (6.3) | 13.0 (6.4)
Statistical Analysis 1: Comparison: Vertebroplasty vs Control Group; Between group comparisons, confidence intervals, and P values were calculated with the use of analysis-of-covariance models with adjustment for study group assignment, baseline value of the outcome measure, and study center. Negative treatment effects favor the control procedure, and positive treatment effects favor vertebroplasty; Test type: Superiority or Other; p = 0.49, ANCOVA; Adjusted treatment effect = 0.7, 95% CI 2-sided [-1.3 to 2.8]

2. Secondary Outcome: Patient Well-being at 1 Month
Description: Patient well-being was quantified by these tools: Health status outcome using Medical Outcomes Study 36-Item Short-Form General Health Survey (SF-36). Scores on the Medical Outcomes Study 36-Item Short-Form General Health Survey (SF-36), version 2. Subjects completed the SF-36 which consists of 8 sub-scales which are additionally summarized into 2 summary components (physical and mental). The subscales and the summary scales both range from 0 to 100, with (0 = worst imaginable, 100 = best imaginable).
  Pain Frequency Index, Pain Bothersome Index (scores range from 0-4, higher scores indicating more severe pain).
  European Quality of Life (QOL) 5 Dimensions (EQ-5D), scale range -0.1 to 1.0; higher scores indicating a better QOL.
  Study of Osteoporotic Fractures-Activities of Daily Living (SOF ADL6) range from 0 to 18; higher scores = more back-related disability.
Time Frame: Month 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vertebroplasty | Control Group
Number analyzed (Participants) | 67 | 61
units on a scale
  SF-36 summary physical component | 29.7 (9.6) | 28.7 (8.0)
  SF-36 summary mental component | 46.9 (12.0) | 45.6 (14.8)
  Pain frequency index score | 2.1 (1.2) | 2.3 (1.1)
  Pain bothersome index score | 1.9 (1.1) | 2.1 (1.1)
  EQ-5D score | 0.70 (0.18) | 0.64 (0.20)
  SOF-ADL score | 7.7 (3.7) | 8.2 (3.6)
Statistical Analysis 1: Comparison: Vertebroplasty vs Control Group; SF-36 Physical Component Summary treatment effect; Test type: Superiority or Other; p = 0.45, ANCOVA; Treatment Effect = 1.0, 95% CI 2-sided [-1.7 to 3.7]
Statistical Analysis 2: Comparison: Vertebroplasty vs Control Group; SF-36 Mental Component Summary treatment effect; Test type: Superiority or Other; p = 0.83, ANCOVA; Treatment Effect = 1.0, 95% CI 2-sided [-3.7 to 4.6]
Statistical Analysis 3: Comparison: Vertebroplasty vs Control Group; Pain Frequency Index treatment effect; Test type: Superiority or Other; p = 0.33, ANCOVA; Treatment Effect = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 4: Comparison: Vertebroplasty vs Control Group; Pain Bothersome Index treatment effect; Test type: Superiority or Other; p = 0.33, ANCOVA; Treatment Effect = 0.33, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 5: Comparison: Vertebroplasty vs Control Group; EQ-5D Index treatment effect; Test type: Superiority or Other; p = 0.13, ANCOVA; Treatment Effect = 0.05, 95% CI 2-sided [-0.01 to 0.11]
Statistical Analysis 6: Comparison: Vertebroplasty vs Control Group; SOF-ADL treatment effect; Test type: Superiority or Other; p = 0.5, ANCOVA; Treatment Effect = 0.4, 95% CI 2-sided [-0.8 to 1.6]

3. Primary Outcome: Patient's Rating of Average Pain at 1 Month
Description: Patient's rating of average pain intensity during the preceding 24 hours at 1 month. The rating scale was from 0 to 10, with higher scores indicating more severe pain.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vertebroplasty | Control Group
Number analyzed (Participants) | 67 | 61
units on a scale | 3.9 (2.9) | 4.6 (3.0)
Statistical Analysis 1: Comparison: Vertebroplasty vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.19, ANCOVA; Adjusted treatment effect = 0.7, 95% CI 2-sided [-0.3 to 1.7]

ADVERSE EVENTS:
Time Frame: 12 months from baseline
Arm/Group | Vertebroplasty | Control Group
Serious Adverse Events (participants affected / at risk) | 1/68 | 1/61
Other Adverse Events (participants affected / at risk) | 0/68 | 0/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vertebroplasty (N=68) | Control Group (N=61)
Surgical injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — One participant in the vertebroplasty group had an injury to the thecal sac during the procedure resulting in hospitalization.
Tachycardia and rigors (Cardiac disorders) | 0 (0) | 1 (1) — One patient in the control group was hospitalized overnight after the procedure with tachycardia and rigors of unknown cause

LIMITATIONS AND CAVEATS:
The possible role of the placebo effect on outcomes remains unclear. Crossover at 1 month was allowed, which complicated the interpretation of between-group outcome differences. Other medical treatments received were not compared to study groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No